CLINICAL TRIAL: NCT04163445
Title: Comparison of Different TKAs Using Objective Dynamic Functional Analysis
Brief Title: Comparison of TKAs Using Force Plate Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russell Nevins, M.D. (Other)
Collaborators: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Russell Nevins, M.D., Chief of Surgery, Desert Orthopedic Center
Organization: Desert Orthopedic Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17IISK01 0
Record Dates: First submitted 2019-11-06; First posted 2019-11-14 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty; Knee Injuries; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patient will be randomized to one of 2 treatment arms using a random number generator. The care provider will not be blinded as he will be implanting the device and following the patients' progress in clinic postoperatively, including radiographs which will show the implants. He will be blinded, however, to the results of the KOOS score and the data derived from the force plate analysis. The research assistants performing those assessments will be blinded to which treatment arm the patient belongs to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Depuy Attune (Active Comparator): Subjects will have been implanted with the Depuy Attune PCR TKA
  Interventions: Device: Depuy Synthes ATTUNE PCR TKA
- MicroPort Medial Pivot (Active Comparator): Subjects will have been implanted with the Microport Evolution Medial Pivot TKA
  Interventions: Device: MicroPort Orthopedics EVOLUTION Medial Pivot TKA

INTERVENTIONS:
Device: MicroPort Orthopedics EVOLUTION Medial Pivot TKA — Subjects will have been implanted with the Microport Evolution Medial Pivot TKA
  Arms: MicroPort Medial Pivot
Device: Depuy Synthes ATTUNE PCR TKA — Subjects will have been implanted with the Depuy Attune PCR TKA
  Arms: Depuy Attune

SUMMARY:
The purpose of this study is to evaluate performance of two modern total knee arthroplasty designs using patient reported outcomes and force exhibited during various activities of daily living.

DETAILED DESCRIPTION:
48 patients with primary osteoarthritis of the knee who have been appropriately designated for treatment with a total knee arthroplasty (TKA) will be randomly assigned to one of two groups; one group (24 patients) will receive a Depuy Attune PCR knee implant, and one group (24 patients) will receive a MicroPort Orthopedics Evolution Medial Pivot knee implant utilizing standard and modern techniques. These two implants are designed to recreate the kinematic motion of a native knee articulation using different biomechanical design philosophies.

The patients will be monitored post-operatively using subjective and objective measures. Subjective patient reported outcomes will be analyzed using the Knee Injury and Osteoarthritis Outcome Score (KOOS), recorded preoperatively, as well as at 6 weeks, and 3 months postoperatively. Objective outcomes will be measured by having the patients perform four activities over force plates that will measure the amount of force a patient generates. The four activities will be: walking, standing from a seated position in a chair, squatting to a seated position, and walking up stairs. These objective measures will also be recorded preoperatively, 6 weeks, and 3 months postoperatively. The patient reported outcomes and the objective measures will then be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been appropriately designated for treatment with a primary total knee arthroplasty
* Subjects who are willing to participate and are willing to sign the Informed Consent/HIPPA documents.

Exclusion Criteria:

* Subjects who are unsuitable candidates for the two types of knee implants under investigation.
* Subjects with significant deformities or arthritis that might affect the procedural decision making, expected outcomes and functions are total knee arthroplasty.
* Subjects with significant comorbidities that might be at an increased risk of post-operative complications.
* Subjects who are unwilling to sign Informed Consent/HIPAA documents.
* Subjects who cannot perform the required activities after the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | pre-operatively
  KOOS Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms
Knee Injury and Osteoarthritis Outcome Score | 6 weeks post-operatively
  KOOS Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms
Knee Injury and Osteoarthritis Outcome Score | 3 months post-operatively
  KOOS Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms
Force generated by operative extremity - walking | pre-operatively
  Distribution of maximum force between implanted and non- implanted leg during walking
Force generated by operative extremity - walking | 6 weeks post-operatively
  Distribution of maximum force between implanted and non- implanted leg during walking
Force generated by operative extremity - walking | 3 months post-operatively
  Distribution of maximum force between implanted and non- implanted leg during walking
Force generated by operative extremity - standing from seated position | pre-operatively
  Distribution of maximum force between implanted and non- implanted leg during standing from a seated position in a chair
Force generated by operative extremity - standing from seated position | 6 weeks post-operatively
  Distribution of maximum force between implanted and non- implanted leg during standing from a seated position in a chair
Force generated by operative extremity - standing from seated position | 3 months post-operatively
  Distribution of maximum force between implanted and non- implanted leg during standing from a seated position in a chair
Force generated by operative extremity - squatting to a seated position | pre-operatively
  Distribution of maximum force between implanted and non- implanted leg during squatting to a seated position
Force generated by operative extremity - squatting to a seated position | 6 weeks post-operatively
  Distribution of maximum force between implanted and non- implanted leg during squatting to a seated position
Force generated by operative extremity - squatting to a seated position | 3 months post-operatively
  Distribution of maximum force between implanted and non- implanted leg during squatting to a seated position
Force generated by operative extremity - walking up stairs | pre-operatively
  Distribution of maximum force between implanted and non- implanted leg during walking up stairs
Force generated by operative extremity - walking up stairs | 6 weeks post-operatively
  Distribution of maximum force between implanted and non- implanted leg during walking up stairs
Force generated by operative extremity - walking up stairs | 3 months post-operatively
  Distribution of maximum force between implanted and non- implanted leg during walking up stairs

CONTACTS AND LOCATIONS:
Overall Officials: Russell Nevins, Principal Investigator — Desert Orthopedics
Locations (1):
- Desert Orthopaedic Center, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No